CLINICAL TRIAL: NCT06317870
Title: Pericapsular Nerve Block Versus Intrathecal Morphine for Analgesia After Primary Hip Arthroplasty: a Double Blind, Non-inferiority Study
Brief Title: Pericapsular Nerve Block Versus Intrathecal Morphine for Analgesia After Primary Hip Arthroplasty
Acronym: PENGIT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Principal Investigator, Eric Albrecht, Prof. Dr. Med. Eric Albrecht, Associate Professor, University of Lausanne, Centre Hospitalier Universitaire Vaudois
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CHUV_PENGIT
Record Dates: First submitted 2024-03-04; First posted 2024-03-19 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Analgesia; Hip Arthropathy; Post Operative Pain
Keywords: nerve block; intrathecal morphine; postoperative pain; hip arthroplasty
MeSH Terms: conditions — Agnosia; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: single centered, prospective, double blinded non inferiority trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: quadruple
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PENG group (Experimental): Pericapsular nerve group block
  Interventions: Procedure: Pericapsular nerve group block (PENG)
- ITM group (Active Comparator): intrathecal morphine injection
  Interventions: Procedure: Intrathecal morphine

INTERVENTIONS:
Procedure: Intrathecal morphine — Spinal anesthesia will be performed as follows: patient will be placed in the lateral decubitus position on the non-operative side. Using sterile gloves red chlorhexidine 2% alcohol solution will be used for skin disinfection. The site will be secured with a sterile drape, and the L4-L5 lumbar space identified. After subcutaneous local infiltration with 1% lidocaine, a 25G Whitacre pencil point spinal needle will be used to access the intrathecal space with free flow of cerebrospinal fluid as confirmation. A mixture of 12.5 mg of isobaric bupivacaine and 100 mcg of morphine will be administered intrathecally.
  After the spinal anesthesia, the intrathecal morphine (ITM) group will receive a sham PENG block with the block needle inserted subcutaneously, the anesthesiologist using the same verbal block confirmation commands "aspirate, inject" but the needle withdrawn without injection. This will create the appearance of an identical cutaneous injection site to ensure patient blinding.
  Arms: ITM group
Procedure: Pericapsular nerve group block (PENG) — Spinal anesthesia with intrathecal injection of 12.5 mg of isobaric bupivacaine will be performed, followed by a PENG block.
  After skin disinfection, a low frequency curvilinear ultrasound probe (2-5 MHz 8870, BK ultrasound, Peabody Massachussets, US) with a sterile covering will be used to identify the anterior inferior iliac spine, the pubic eminence and the psoas tendon with its fascial plane. A 22 gauge 10cm block needle (Sonoplex® Pajunk, Geisingen, DE), will be used to enter the fascial plane and 20ml of 0.75% Ropivacain (Fresenius Kabi, Krienz CH) will be injected.
  Arms: PENG group

SUMMARY:
The aim of this clinical trial is to compare the analgesic effect of pericapsular nerve block (PENG) with intrathecal morphine in patients scheduled for total hip replacement surgery. The main question to be answered is whether the PENG block is equivalent to intrathecal morphine in reducing postoperative pain.

Participants will be randomised into two groups. Patients assigned to the PENG group will receive spinal anaesthesia with local anaesthetic (isobaric bupivacaine) alone and a PENG block. Patients assigned to the intrathecal morphine (ITM) group will receive spinal anaesthesia with a mixture of local anaesthetic (isobaric bupivacaine) and morphine (100 mcg) and a sham PENG block to ensure patient blinding.

DETAILED DESCRIPTION:
The aim of this double-blind, non-inferiority study is to compare the analgesic effect of a PENG block with intrathecal morphine in patients scheduled for total hip arthroplasty. Postoperative morphine consumption and pain scores, morphine-related adverse effects and functional parameters will be compared between two groups.

The investigators believe that PENG block provides postoperative analgesia equivalent to intrathecal morphine. The research team plans to enrol 80 patients and randomise them to two groups - pericapsular nerve block (PENG) or intrathecal morphine (ITM). After written informed consent, patients will be allocated to one of the two groups according to a computer-generated randomisation list. The PENG group will receive central spinal anaesthesia with 12.5 mg isobaric bupivacaine followed by a PENG block with 20 cc of 0.75% ropivacaine. ITM groups will receive central spinal anaesthesia with 12.5 mg isobaric bupivacaine and 100 mcg morphine followed by a sham PENG block.

During the surgery, 0.15 mg/kg of dexamethasone iv, 1g acetaminophen iv, 30mg ketorolac iv and 40mg/kg magnesium iv will be administered for post operative analgesia.

In the post-operative care unit, pain management will be provided with as needed with 2mg of IV morphine at ten minute intervals for pain scores >3. Once spinal motor block has ceded, the patients will be transferred to the surgical ward with a morphine patient controlled analgesia (PCA) pump. The pump parameters will allow 2 mg boluses of morphine with a 10-minute lockout and a maximum dose of 40 mg in 4 hours. Basal analgesia will be provided with paracetamol (1g/6h) and ibuprofen (400mg/8h). Ondansetron (4mg IV) will be provided in case of nausea or vomiting. A research assistant will conduct post operative visits at 2h, 1 day and 2 days post-operatively to record research data. Functional testing will be performed at day 1 and 2 by physiotherapy personnel.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* ASA (American Society of Anaesthesiologists) I-III
* 18 years of age or older
* Patients scheduled for elective primary hip arthroplasty
* Able to give written conformed consent autonomously

Exclusion Criteria:

* Refusal or inability to give consent
* Allergy to any of: ropivacaine, paracetamol, ibuprofen, ketorolac, morphine, ondansetron or dexamethasone
* Bleeding diathesis
* Neurological deficit of the operative side
* Existing preoperative opioid use
* Renal insufficiency (GFR<30ml/min according to the Cockroft-Gault formula)
* Hepatic insufficiency
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-09-10 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative postoperative morphine consumption at day 1 | 24 hours postoperatively
  total consumption in mg

SECONDARY OUTCOMES:
Morphine consumption in the recovery room | from admission till discharge from the recovery room, up to 2 hours
  consumption in mg
PCA administered morphine consumption at day 2 | at day 2 postoperatively
  consumption in mg administered by PCA
rest and dynamic pain scores | at 2 hours, day 1 and day 2 postoperatively
  Visual Analogue Scale(VAS), 0-10
Incidence of postoperative nausea and vomiting | at 2 hours, day 1 and day 2 postoperatively
  Presence of nausea or vomiting in the postoperative period
Incidence of pruritus | at 2 hours, day 1 and day 2 postoperatively
  Presence of pruritus in the postoperative period
Incidence of urinary retention requiring bladder catheterisation | from surgery till day 2 postoperatively
  Urinary retention requiring catheterisation
Duration of analgesia | from the time the study procedure is performed up to 36 hours after surgery
  Time between study procedure and the first dose of iv morphine
operated limb quadriceps strength | at day 1 and day 2 postoperatively
  Medical Research Council Manual Muscle Testing scale, 0-5
Walking test | at day 1 and 2 postoperatively
  maximum distance travelled (meters)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Lausanne, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anger M, Valovska T, Beloeil H, Lirk P, Joshi GP, Van de Velde M, Raeder J; PROSPECT Working Group* and the European Society of Regional Anaesthesia and Pain Therapy. PROSPECT guideline for total hip arthroplasty: a systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2021 Aug;76(8):1082-1097. doi: 10.1111/anae.15498. Epub 2021 May 20. PMID 34015859
- [Background] Gonvers E, El-Boghdadly K, Grape S, Albrecht E. Efficacy and safety of intrathecal morphine for analgesia after lower joint arthroplasty: a systematic review and meta-analysis with meta-regression and trial sequential analysis. Anaesthesia. 2021 Dec;76(12):1648-1658. doi: 10.1111/anae.15569. Epub 2021 Aug 27. PMID 34448492
- [Background] Vitola E, Buraka N, Erts R, Golubovska I, Miscuks A. Effect of different low doses of intrathecal morphine (0.1 and 0.2 mg) on pain and vital functions in patients undergoing total hip arthroplasty: a randomised controlled study. BMC Anesthesiol. 2022 Dec 5;22(1):377. doi: 10.1186/s12871-022-01919-8. PMID 36471258
- [Background] Kuchalik J, Granath B, Ljunggren A, Magnuson A, Lundin A, Gupta A. Postoperative pain relief after total hip arthroplasty: a randomized, double-blind comparison between intrathecal morphine and local infiltration analgesia. Br J Anaesth. 2013 Nov;111(5):793-9. doi: 10.1093/bja/aet248. Epub 2013 Jul 19. PMID 23872462
- [Background] Souron V, Delaunay L, Schifrine P. Intrathecal morphine provides better postoperative analgesia than psoas compartment block after primary hip arthroplasty. Can J Anaesth. 2003 Jun-Jul;50(6):574-9. doi: 10.1007/BF03018643. PMID 12826549
- [Background] Kearns R, Macfarlane A, Grant A, Puxty K, Harrison P, Shaw M, Anderson K, Kinsella J. A randomised, controlled, double blind, non-inferiority trial of ultrasound-guided fascia iliaca block vs. spinal morphine for analgesia after primary hip arthroplasty. Anaesthesia. 2016 Dec;71(12):1431-1440. doi: 10.1111/anae.13620. Epub 2016 Oct 7. PMID 27714758
- [Background] Roofthooft E, Joshi GP, Rawal N, Van de Velde M; PROSPECT Working Group* of the European Society of Regional Anaesthesia and Pain Therapy and supported by the Obstetric Anaesthetists' Association. PROSPECT guideline for elective caesarean section: updated systematic review and procedure-specific postoperative pain management recommendations. Anaesthesia. 2021 May;76(5):665-680. doi: 10.1111/anae.15339. Epub 2020 Dec 28. PMID 33370462
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Pascarella G, Costa F, Del Buono R, Pulitano R, Strumia A, Piliego C, De Quattro E, Cataldo R, Agro FE, Carassiti M; collaborators. Impact of the pericapsular nerve group (PENG) block on postoperative analgesia and functional recovery following total hip arthroplasty: a randomised, observer-masked, controlled trial. Anaesthesia. 2021 Nov;76(11):1492-1498. doi: 10.1111/anae.15536. Epub 2021 Jul 1. PMID 34196965
- [Background] Lin DY, Brown B, Morrison C, Fraser NS, Chooi CSL, Cehic MG, McLeod DH, Henningsen MD, Sladojevic N, Kroon HM, Jaarsma RL. The Pericapsular Nerve Group (PENG) block combined with Local Infiltration Analgesia (LIA) compared to placebo and LIA in hip arthroplasty surgery: a multi-center double-blinded randomized-controlled trial. BMC Anesthesiol. 2022 Aug 6;22(1):252. doi: 10.1186/s12871-022-01787-2. PMID 35933328
- [Background] Hu J, Wang Q, Hu J, Kang P, Yang J. Efficacy of Ultrasound-Guided Pericapsular Nerve Group (PENG) Block Combined With Local Infiltration Analgesia on Postoperative Pain After Total Hip Arthroplasty: A Prospective, Double-Blind, Randomized Controlled Trial. J Arthroplasty. 2023 Jun;38(6):1096-1103. doi: 10.1016/j.arth.2022.12.023. Epub 2022 Dec 16. PMID 36529195
- [Background] Aliste J, Layera S, Bravo D, Jara A, Munoz G, Barrientos C, Wulf R, Branez J, Finlayson RJ, Tran Q. Randomized comparison between pericapsular nerve group (PENG) block and suprainguinal fascia iliaca block for total hip arthroplasty. Reg Anesth Pain Med. 2021 Oct;46(10):874-878. doi: 10.1136/rapm-2021-102997. Epub 2021 Jul 20. PMID 34290085